CLINICAL TRIAL: NCT03622333
Title: Clinic, Pathologic and Genetic Characterization of Patients With Familial Carcinoid Tumors (Study From the GTE, Groupe d'étude Des Tumeurs Endocrines)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PO18020
Record Dates: First submitted 2018-02-22; First posted 2018-08-09 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-02

CONDITIONS: Small Intestinal Carcinoid Tumors
Keywords: Neuroendocrine tumors; carcinoid tumors; midgut; small intestine; genetic predisposition; hereditary
MeSH Terms: conditions — Neuroendocrine Tumors; Carcinoid Tumor; Genetic Predisposition to Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Familial Carcinoid Tumors (Experimental): All patients with proven Familial Carcinoid Tumors
  Interventions: Genetic: Research of constitutional genetic alterations

INTERVENTIONS:
Genetic: Research of constitutional genetic alterations — Tumor DNA extraction Blood sample and constitutional DNA extraction CGH-array, Exome sequencing Bio-informatic analysis

SUMMARY:
Small intestine carcinoid tumors are rare. Small intestine Familial Carcinoid Tumors (FCT) are defined by the occurrence of at least 2 cases of this tumor type in first- or second-degree relatives. The estimated prevalence of FCT is 2.6%-3.7% in patients with small intestine carcinoid tumors. Because of its rarity, epidemiologic, clinic and pathologic features of FCT have been scarcely described. Molecular abnormalities associated with FCT have been poorly explored. Constitutional genetic factors predisposing to FCT have not been discovered to date. Only one abnormality (mutation of the IPMK gene) has been reported in one FCT family only, but not found in other series.

The main objective of this study is to identify the constitutional factors predisposing to small-intestine FCT (and other midgut localizations: ascending colon and appendix). The secondary objectives are to describe the clinic and pathologic features associated with FCT.

ELIGIBILITY:
inclusion criteria :

* Small-intestine (or ascending colon or appendix) neuroendocrine tumor (proven histologically)
* At least one first- or second-degree relative with a small-intestine (or ascending colon or appendix) neuroendocrine tumor (proven histologically)
* Agreement to participate to the study exclusion criteria :
* Subjects unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-05-28 (Actual); Primary Completion 2022-05-28 (Estimated); Study Completion 2022-11-28 (Estimated)

PRIMARY OUTCOMES:
Deletion | day 0
  Quantitative Constitutional genetic alterations detected by comparative genomic hybridization (CGH array)
duplication | Day 0
  Quantitative Constitutional genetic alterations detected by comparative genomic hybridization (CGH array)
amplification | Day 0
  Quantitative Constitutional genetic alterations detected by comparative genomic hybridization (CGH array)
mutation | Day 0
  qualitative Constitutional genetic alterations detected by NGS (Next Generation Sequencing)

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France